CLINICAL TRIAL: NCT03756675
Title: Haploidentical Peripheral Blood Stem Cell Transplantation for Acute Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Supervisor of Hematology, Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: Haplo-PBSCT for AL
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Acute Leukemia
Keywords: allogeneic stem cell transplantation; G-CSF-mobilized peripheral blood stem cell; haplotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- haplotype PBSCT group: Subjects in this group will receive haplotype peripheral blood stem cell transplantation (PBSCT) of "GIAC" system in the treatment of acute leukemia.
  Interventions: Other: haplotype PBSCT

INTERVENTIONS:
Other: haplotype PBSCT — haplotype peripheral blood stem cell transplantation (PBSCT) of "GIAC" system

SUMMARY:
Allogeneic stem cell transplantation (Allo-HSCT) is the effective and even the only treatment for hematological malignancies. The "GIAC" protocol established by our center has successfully crossed the HLA barrier in HLA-mismatched/haploidentical HSCT. The protocol entails the following: treating donors with granulocyte colony-stimulating factor (G-CSF) to induce donor immune tolerance, intensified immunologic suppression to both promote engraftment and to prevent GVHD, antithymocyte globulin (ATG) was included for the prophylaxis of GVHD and graft rejection, and combination of G-CSF-primed bone marrow harvest (G-BM) and G-CSF-mobilized peripheral blood stem cell harvest (G-PB) as the source of stem cell grafts. But peripheral blood transplantation is still prevalent. Compared with BM, G-PB is more convenient to collect, and the number of T lymphocytes and CD34+ cells is higher. It is reported that G-PB has a higher implantation rate and even a higher disease-free survival rate in sibiling-identical transplantation compared with BM transplantation, whereas there were also reports with different conclusions. This prospective, one-arm clinical cohort study aims to evaluate the safety and efficacy of haplotype peripheral blood stem cell transplantation (PBSCT) in the treatment of acute leukemia.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (Allo-HSCT) is the effective and even the only treatment for hematological malignancies. The "GIAC" protocol established by our center has successfully crossed the HLA barrier in HLA-mismatched/haploidentical HSCT. The protocol entails the following: treating donors with granulocyte colony-stimulating factor (G-CSF) to induce donor immune tolerance, intensified immunologic suppression to both promote engraftment and to prevent GVHD, antithymocyte globulin (ATG) was included for the prophylaxis of GVHD and graft rejection, and combination of G-CSF-primed bone marrow harvest (G-BM) and G-CSF-mobilized peripheral blood stem cell harvest (G-PB) as the source of stem cell grafts. But peripheral blood transplantation is still prevalent. Compared with BM, G-PB is more convenient to collect, and the number of T lymphocytes and CD34+ cells is higher. It is reported that G-PB has a higher implantation rate and even a higher disease-free survival rate in sibiling-identical transplantation compared with BM transplantation, whereas there were also reports with different conclusions. This prospective, one-arm clinical cohort study aims to evaluate the safety and efficacy of haplotype peripheral blood stem cell transplantation (PBSCT) in the treatment of acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* 2-60 years old, all genders;
* the first complete remission phase (CR1) of acute leukemia;
* planning to receive haplotype PBSCT;
* no uncontrolled current infections (new infections, body temperature still above 38 ℃ after treatment with broad-spectrum antibiotics for 72h, except for other non-infectious factors);
* no organ failure.

Exclusion Criteria:

* with poor compliance;
* with uncontrolled current infections；
* pregnancy;
* donors with contraindications of mobilization and collection of peripheral blood stem cells;
* with mental sickness

Ages: 2 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients aged 2-60, who plan to receive haplotype PBSCT in the first complete remission phase (CR1) of acute leukemia, and with no uncontrolled current infections or organ failure.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
engraftment rate | one year after transplantation
  Neutrophil recovery was defined as an absolute neutrophil count(ANC) of 0.5×10^9/L or more for three consecutive days and platelet recovery, as 20×10^9/L or more for seven consecutive days without transfusion.

SECONDARY OUTCOMES:
cumulative incidence of acute graft-versus-host disease(GVHD) | one year after transplantation
  cumulative incidence of acute graft-versus-host disease(GVHD)
cumulative incidence of chronic GVHD at one year | one year after transplantation
  cumulative incidence of chronic GVHD at one year
cumulative incidence of relapse at one year | one year after transplantation
  Cumulative incidence of relapse was defined as the cumulative incidences of presence of morphological evidence of disease in samples from peripheral blood, bone marrow, or extramedullary sites, or by the recurrence and sustained presence of pre-transplantation chromosomal abnormalities.
cumulative incidence of non-relapse mortality (NRM) at one year | one year after transplantation
  NRM was defined as the death without disease progression or relapse.
overall survival at one year | one year after transplantation
  OS was defined as the time from the date of first dose until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shen MZ, Hong SD, Lou R, Chen RZ, Zhang XH, Xu LP, Wang Y, Yan CH, Chen H, Chen YH, Han W, Wang FR, Wang JZ, Liu KY, Huang XJ, Mo XD. A comprehensive model to predict severe acute graft-versus-host disease in acute leukemia patients after haploidentical hematopoietic stem cell transplantation. Exp Hematol Oncol. 2022 May 3;11(1):25. doi: 10.1186/s40164-022-00278-x. PMID 35505384
- [Derived] Shen MZ, Hong SD, Wang J, Zhang XH, Xu LP, Wang Y, Yan CH, Chen H, Chen YH, Han W, Wang FR, Wang JZ, Liu KY, Huang XJ, Mo XD. A Predicted Model for Refractory/Recurrent Cytomegalovirus Infection in Acute Leukemia Patients After Haploidentical Hematopoietic Stem Cell Transplantation. Front Cell Infect Microbiol. 2022 Mar 22;12:862526. doi: 10.3389/fcimb.2022.862526. eCollection 2022. PMID 35392613
- [Derived] Ma YR, Zhang X, Xu L, Wang Y, Yan C, Chen H, Chen Y, Han W, Wang F, Wang J, Liu K, Huang X, Mo X. G-CSF-Primed Peripheral Blood Stem Cell Haploidentical Transplantation Could Achieve Satisfactory Clinical Outcomes for Acute Leukemia Patients in the First Complete Remission: A Registered Study. Front Oncol. 2021 Mar 15;11:631625. doi: 10.3389/fonc.2021.631625. eCollection 2021. PMID 33791217